CLINICAL TRIAL: NCT00045903
Title: CBT Augmentation for SRI Pharmacotherapy in OCD
Brief Title: Cognitive Behavioral Therapy Plus Drug Treatment for Obsessive Compulsive Disorder
Acronym: Aug1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #4734R; R01MH045436-01 (NIH); DSIR AT-CT
Record Dates: First submitted 2002-09-13; First posted 2002-09-17 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2012-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exposure and Ritual Prevention (Experimental): Exposure and Ritual Prevention Therapy
  Interventions: Behavioral: Exposure and Ritual Prevention (Cognitive Behavioral Therapy)
- Stress Management (Active Comparator): Stress Management Therapy
  Interventions: Behavioral: Stress Management Therapy (Cognitive Behavior Therapy)

INTERVENTIONS:
Behavioral: Exposure and Ritual Prevention (Cognitive Behavioral Therapy)
  Arms: Exposure and Ritual Prevention
Behavioral: Stress Management Therapy (Cognitive Behavior Therapy)
  Arms: Stress Management

SUMMARY:
This study will evaluate the effectiveness of two cognitive behavioral therapies (CBTs) in treating obsessive compulsive disorder (OCD) in patients who are taking medication but still have residual symptoms.

DETAILED DESCRIPTION:
Participants remain on their current OCD medication and are randomly assigned to receive one of two CBTs: exposure and ritual prevention or stress management therapy. Exposure and ritual prevention involves imaginal and in-vivo exposure and requires that participants refrain from ritualizing. Stress management involves relaxation, assertiveness training, and structured problem-solving. Therapy occurs twice per week for 2 months. Participants are assessed verbally by an independent evaluator and are asked to complete self-rating forms. Patients who respond are followed for up to 1 additional year. Participants continue to take the same medication and the same monthly therapy for the first 6 months of follow-up. During the second 6 months of follow-up, participants discontinue therapy but continue taking the same medication.

For information on a related study, please follow this link:

http://clinicaltrials.gov/show/NCT00389493

ELIGIBILITY:
Inclusion Criteria:

* Obsessive-Compulsive Disorder (OCD) diagnosis
* Currently taking a serotonin reuptake inhibitor (SRI, i.e. clomipramine, fluoxetine, fluvoxamine, paroxetine, sertraline, or citalopram) for OCD

Exclusion Criteria:

* Medical or psychiatric conditions that would make participation in the study hazardous
* Intensive cognitive-behavioral therapy while on an adequate dose and duration of an SRI for OCD

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2000-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms measured at Month 2 | 2 months

SECONDARY OUTCOMES:
General functioning measured at Month 2 | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Liebowitz, MD, Principal Investigator — New York State Psychiatric Institute; Edna Foa, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - New York State Psychiactic Institute, Anxiety Disorders Clinic, New York, New York
  - University of Pennsylvania Center for the Treatment and Study of Anxiety, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Farris SG, McLean CP, Van Meter PE, Simpson HB, Foa EB. Treatment response, symptom remission, and wellness in obsessive-compulsive disorder. J Clin Psychiatry. 2013 Jul;74(7):685-90. doi: 10.4088/JCP.12m07789. PMID 23945445
- [Derived] Foa EB, Simpson HB, Liebowitz MR, Powers MB, Rosenfield D, Cahill SP, Campeas R, Franklin M, Hahn CG, Hembree EA, Huppert JD, Schmidt AB, Vermes D, Williams MT. Six-month follow-up of a randomized controlled trial augmenting serotonin reuptake inhibitor treatment with exposure and ritual prevention for obsessive-compulsive disorder. J Clin Psychiatry. 2013 May;74(5):464-9. doi: 10.4088/JCP.12m08017. PMID 23759449